CLINICAL TRIAL: NCT02344745
Title: The Use of Lavender Aromatherapy to Decrease Women's Anxiety and Perception of Pain During Multi-channel Urodynamics Procedure
Brief Title: Lavender Aromatherapy for Anxiety During Urodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Begum Ozel, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-14-00444
Record Dates: First submitted 2015-01-07; First posted 2015-01-26 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Anxiety; Pain
Keywords: Lavender; Aromatherapy; Urodynamics
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Distilled water
  Interventions: Other: Distilled water
- Lavender (Experimental): Lavandula angustifolia essential oil (Aura Cacia)
  Interventions: Other: Lavandula angustifolia essential oil (Aura Cacia)

INTERVENTIONS:
Other: Lavandula angustifolia essential oil (Aura Cacia) — The participants will be instructed to take a deep breath while holding the towel with two drops of essential oil 3 inches from her face before the start of the procedure and will be instructed to continue to take normal breaths subsequently during the procedure.
  Arms: Lavender
Other: Distilled water — The participants will be instructed to take a deep breath while holding the towel with two drops of distilled water 3 inches from her face before the start of the procedure and will be instructed to continue to take normal breaths subsequently during the procedure.
  Arms: Control

SUMMARY:
Urodynamics are performed in the evaluation of urinary incontinence in women considering surgery or who have failed conservative therapies. Urodynamic testing requires the placement of small catheters into the bladder and the vagina or rectum. Many women experience anxiety around the procedure which can affect patient satisfaction. Lavender aromatherapy has been associated with decreased anxiety in a variety of clinical situations. The purpose of this study is to determine a difference in self-reported anxiety and pain levels before, during, and after multichannel urodynamics in patients given lavender aromatherapy versus placebo. This study design is a randomized control trial. Women scheduled for urodynamic testing at the Los Angeles County University of Southern California (LAC+USC) Urogynecology clinic will be invited to participate. Participants will be randomized to the aromatherapy or the placebo group after informed consent is obtained and immediately before undergoing multichannel urodynamics. The participants will complete the Hospital Anxiety and Depression Survey (HADS) at baseline. They will be asked to rate their level of anxiety and pain before, during, and 15 min after the study using the visual analogue scale and Wong-Baker pain scale. At the end the participants will also be asked to rate their satisfaction with the visit overall. The primary endpoint is defined as anxiety immediately after catheters are placed. Data will be entered into a coded database for analysis using the independent samples t test, the Mann-Whitney U test, and the chi square test. Intention to treat analysis will be used.

DETAILED DESCRIPTION:
This study design is a randomized placebo control trial.

Aside from randomization to aromatherapy versus placebo, no procedures will be performed for study purposes that would not be normally performed in the clinical evaluation.

Women scheduled for urodynamic testing at the Los Angeles County University of Southern California (LAC+USC) Urogynecology clinic will be invited to participate. Participants who meet inclusion criteria will be randomized to the aromatherapy or the placebo group after informed consent is obtained and immediately before undergoing multichannel urodynamics. Sequentially numbered sealed opaque envelopes containing the identity of the study arm will be used for randomization. The urogynecology clinic nurse will prepare the aromatherapy versus distilled water on the paper towel that the patient is routinely given to hold over their mouths when asked to cough during the procedure; two drops of each will be utilized. Before the physician comes in, the nurse will ask the participant to take a deep breath while holding the towel 3 inches from her face and will instruct the participant to continue to take normal breaths subsequently. It will not be possible to blind the participants or the examiner to the assigned group since the lavender oil will have a different scent than the placebo. However, the use of distilled water on the towel will allow the possibility that the deep breathing accompanying the instruction may have an effect on reported pain and anxiety.

The participant will undergo the standard clinic exam in standardized order. The participants will complete the Hospital Anxiety and Depression Survey (HADS) at baseline. The HADS is reliable instrument for detecting states of depression and anxiety in the setting of a hospital medical outpatient clinic; it is available in English and Spanish versions. This will be used to establish their baseline anxiety levels. Participants will then be asked to rate their level of anxiety and pain immediately before beginning the exam, immediately after catheter placement, and 15 min after termination of the study using a 10 point visual analogue scale and the Wong-Baker pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over,
* Scheduled to undergo multichannel urodynamic study,
* Able to give informed consent,
* Able to read and write in English or Spanish,
* Anxiety score > 0 on numerical scale at baseline

Exclusion Criteria:

* Any contraindication to multichannel urodynamic study (active urinary tract infection, active pelvic infection, glucosuria, severe hypertension, or any other condition that might be worsened by an uncomfortable test),
* Allergy to lavender oil, or any of its components

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Begum Ozel, M.D., Principal Investigator — University of Southern California
Locations (1):
- Los Angeles Count + USC Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Stea S, Beraudi A, De Pasquale D. Essential oils for complementary treatment of surgical patients: state of the art. Evid Based Complement Alternat Med. 2014;2014:726341. doi: 10.1155/2014/726341. Epub 2014 Feb 24. PMID 24707312
- [Background] Yeung JY, Eschenbacher MA, Pauls RN. Pain and embarrassment associated with urodynamic testing in women. Int Urogynecol J. 2014 May;25(5):645-50. doi: 10.1007/s00192-013-2261-1. Epub 2013 Nov 27. PMID 24280994
- [Background] Yokoyama T, Nozaki K, Nose H, Inoue M, Nishiyama Y, Kumon H. Tolerability and morbidity of urodynamic testing: a questionnaire-based study. Urology. 2005 Jul;66(1):74-6. doi: 10.1016/j.urology.2005.01.027. PMID 15992874
- [Background] Ku JH, Kim SW, Kim HH, Paick JS, Son H, Oh SJ. Patient experience with a urodynamic study: a prospective study in 208 patients. J Urol. 2004 Jun;171(6 Pt 1):2307-10. doi: 10.1097/01.ju.0000125144.82338.0c. PMID 15126810
- [Background] Soltani R, Soheilipour S, Hajhashemi V, Asghari G, Bagheri M, Molavi M. Evaluation of the effect of aromatherapy with lavender essential oil on post-tonsillectomy pain in pediatric patients: a randomized controlled trial. Int J Pediatr Otorhinolaryngol. 2013 Sep;77(9):1579-81. doi: 10.1016/j.ijporl.2013.07.014. Epub 2013 Aug 8. PMID 23932834
- [Background] Muzzarelli L, Force M, Sebold M. Aromatherapy and reducing preprocedural anxiety: A controlled prospective study. Gastroenterol Nurs. 2006 Nov-Dec;29(6):466-71. doi: 10.1097/00001610-200611000-00005. PMID 17273013
- [Background] Grunebaum LD, Murdock J, Castanedo-Tardan MP, Baumann LS. Effects of lavender olfactory input on cosmetic procedures. J Cosmet Dermatol. 2011 Jun;10(2):89-93. doi: 10.1111/j.1473-2165.2011.00554.x. PMID 21649812
- [Background] Braden R, Reichow S, Halm MA. The use of the essential oil lavandin to reduce preoperative anxiety in surgical patients. J Perianesth Nurs. 2009 Dec;24(6):348-55. doi: 10.1016/j.jopan.2009.10.002. PMID 19962101
- [Background] Fayazi S, Babashahi M, Rezaei M. The effect of inhalation aromatherapy on anxiety level of the patients in preoperative period. Iran J Nurs Midwifery Res. 2011 Fall;16(4):278-83. PMID 23449862
- [Background] Olapour A, Behaeen K, Akhondzadeh R, Soltani F, Al Sadat Razavi F, Bekhradi R. The Effect of Inhalation of Aromatherapy Blend containing Lavender Essential Oil on Cesarean Postoperative Pain. Anesth Pain Med. 2013 Summer;3(1):203-7. doi: 10.5812/aapm.9570. Epub 2013 Jul 1. PMID 24223363
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Ozel BZ, Quevedo A, Jung C, Shirazi F, Dancz CE. Lavender Aromatherapy for Anxiety and Pain During Multichannel Urodynamics: A Randomized Controlled Pilot Trial. Female Pelvic Med Reconstr Surg. 2021 Nov 1;27(11):654-658. doi: 10.1097/SPV.0000000000001032. PMID 33626029

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Lavender
Started | 40 | 40
Completed | 38 | 40
Not Completed | 2 | 0
Not completed — Data collection sheets were lost | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Lavender | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (7.5) | 49.0 (8.0) | 48.5 (7.9)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 39 | 76
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Anxiety [Median (Full Range); unit: cm] — Anxiety was measured using a visual analogue scale, from 0-10 cm. All measurements were rounded to the nearest 0.5 cm. Since all participants had baseline anxiety, the lowest score recorded was 1. Higher values indicate more anxiety.
  cm | 4 [1 to 9] | 5 [1 to 10] | 5 [1 to 10]
Pain [Median (Full Range); unit: units on a scale] — Pain was measured on the Wong Baker scale from 0-10. Higher values indicate more pain.
  units on a scale | 0 [0 to 5] | 0 [0 to 4] | 0 [0 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Measured by VAS
Description: Anxiety was measured using a visual analogue scale, from 0-10 cm. All measurements were rounded to the nearest 0.5 cm. Higher values indicate more anxiety.
Time Frame: At the time of catheter placement
Measure: Median (Full Range); unit: cm
Arm/Group | Control | Lavender
Number analyzed (Participants) | 38 | 40
cm | 4 [0 to 9] | 3 [0 to 8]
Statistical Analysis 1: Comparison: Control vs Lavender; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Wong Baker Pain Scale
Description: Pain was measured on the Wong Baker scale from 0-10. Higher values indicate more pain.
Time Frame: At the time of catheter placement
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control | Lavender
Number analyzed (Participants) | 38 | 40
units on a scale | 0 [0 to 5] | 0 [0 to 9]
Statistical Analysis 1: Comparison: Control vs Lavender; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Anxiety Measured by VAS
Description: as for outcome 1
Time Frame: 15 min after removal of the urodynamics catheters
Measure: Median (Full Range); unit: cm
Arm/Group | Control | Lavender
Number analyzed (Participants) | 38 | 39
cm | 0.5 [0 to 5] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Control vs Lavender; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Wong Baker Pain Scale
Description: Pain was measured on the Wong Baker scale from 0-10. Higher values indicate more pain.
Time Frame: 15 min after removal of the urodynamics catheters
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control | Lavender
Number analyzed (Participants) | 38 | 39
units on a scale | 0 [0 to 5] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Control vs Lavender; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The participants were observed for 60 minutes after administration of aromatherapy.
Arm/Group | Control | Lavender
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No